CLINICAL TRIAL: NCT06110507
Title: Chronic Anergic-anhedonic Depression Open Trial
Acronym: CADOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8903
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Depressive Disorder; Treatment-Resistant; Anergic-anhednic; TRD; TRAD; MAOI; dopamine D2 receptor agonists; D2RAG; dopamine-sensitive
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A form of depression called 'dopamine-sensitive anergic-anhedonic syndrome is usually resistant to standard therapies (TRAD). On the other hand, they respond to dopaminergic approaches for which recommendations have been developed: DATA ('Dopaminergic Antidepressant Therapy Algorithm'). These are two stages starting with non-selective monoamineoxidase inhibitors (MAOI) or dopamine D2 receptor agonists (D2RAG) in 'monotherapy' (DATA1) and proposing to combine them in the event of a partial response (DATA2).

The effectiveness of this approach in the management of TRAD has not yet been evaluated in routine care.

The aim of this study is to evaluate the feasibility and effectiveness in routine care of the DATA recommendations in the management of TRAD presenting to a specialized consultation for resistant depression (short and long-term results).

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years old)
* Man or woman
* Patient covered for consultation at the Expert Resistant Depression Center of Alsace (CEDRA) (CHU-Strasbourg branch) for TRAD between 01 January 2013 and 31 March 2023
* Patient not opposing to the reuse of their data for the purposes of this research

Exclusion Criteria:

* Patient having expressed opposition to participating in the study
* Patient under judicial protection
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patient (≥18 years old) covered for consultation at the Expert Resistant Depression Center of Alsace (CEDRA) (CHU-Strasbourg branch) for TRAD between 01 January 2013 and 31 March 2023
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in remission; Remission time; Survival curves for remissions and responses | 3 months after the patient was taken care of at the Strasbourg University Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CENTRE DE NEUROMODULATION NON INVASIVE DE STRASBOURG (CEMNIS) - CHU de Strasbourg - France, Strasbourg, France